CLINICAL TRIAL: NCT01867528
Title: Laparoscopic Versus Open Adhesiolysis for Small Bowel Obstruction - A Multicenter, Prospective, Randomized, Controlled Trial
Brief Title: Comparison of Laparoscopic Surgery Versus Open Surgery in the Treatment of Adhesive Small Bowel Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUCH-95-150513
Record Dates: First submitted 2013-05-26; First posted 2013-06-04 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Adhesive Small Bowel Obstruction

ARMS (2):
- Laparoscopic adhesiolysis (Experimental)
  Interventions: Procedure: Laparoscopic adhesiolysis
- Open adhesiolysis (Active Comparator)
  Interventions: Procedure: Open adhesiolysis

INTERVENTIONS:
Procedure: Laparoscopic adhesiolysis
  Arms: Laparoscopic adhesiolysis
Procedure: Open adhesiolysis
  Arms: Open adhesiolysis

SUMMARY:
Small bowel obstruction is a common reason for surgical admission. Most common reason for small bowel obstruction is adhesions, which account up to 70-80 % of small bowel obstructions. Large proportion of adhesive small bowel obstructions may be treated nonoperatively, but up to 50-60% may need surgical intervention. Current golden standard for surgical intervention is open adhesiolysis. Recently, retrospective studies have provided encouraging results of laparoscopic adhesiolysis for small bowel obstructions. However, no prospective randomized trials have been carried out and retrospective series carries a high risk for patient selection and bias. Although in general laparoscopy has been associated with shortened hospital stay, less pain and reduced mortality, laparoscopic adhesiolysis for small bowel obstruction has been reported to cause iatrogenic small bowel lesions up to 7% of patients. Aim of the study is to compare open adhesiolysis to laparoscopic adhesiolysis. The investigators hypothesis is that laparoscopic adhesiolysis is safe, will shorten the hospital stay, and reduce mortality compared to open approach.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical and computed tomography-diagnosed adhesive small bowel obstruction AND
* Obstruction is not relieved by conservative methods (nasogastric tube, NPO) including Gastrografin is not passed to colon within 8 hours (48-hour conservative treatment without Gastrografin® is allowed if Gastrografin® is contraindicated (e.g. allergy) or not available)

Exclusion Criteria:

* Strong suspicion of strangulation or clinical peritonitis thus indicating an urgent operative intervention
* Earlier confirmed or strongly suspected peritoneal carcinosis
* Earlier confirmed wide diffuse adhesions of abdominal cavity
* Earlier open surgery for endometriosis
* Earlier generalized diffuse peritonitis (not including local peritonitis such as appendicitis)
* Active abdominal malignancy or remission less than 10 years
* Earlier abdominal region radiotherapy
* Earlier obesity surgery
* 3 or more earlier open abdominal operations (not including caesarean section(s))
* Suspicion of other cause for obstruction than adhesions in CT-scan
* Earlier abdominal surgical operation within 30 days
* Earlier surgical operation for aorta or iliac vessels performed through laparotomy
* Crohn's disease
* Anesthesiological contraindication for laparoscopy
* Missing informed consent
* Age less than 18 years or over 95 years
* Pregnancy
* Patient living in institutional care (such as health centre ward), not including retirement homes
* Over 1 week of hospital stay directly prior surgical consultation

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2013-07; Primary Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Post-operative hospital stay (days) | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days

SECONDARY OUTCOMES:
Passage of stools (post-operative days) | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days
Commence of enteral nutrition (post-operative days) | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days
Mortality | 30 days after randomization
Complications, Clavien-Dindo classification | 30 days after randomization
Number of participants with iatrogenic small bowel lesions | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days
Number of participants with readmission(s) | 30 days after randomization
Number of participant with failure to relieve obstruction | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days
Pain scores on the Visual Analog Scale | Postoperative days 1- 7 or till discharge
Length of epidural catheter analgesia (days) | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days
Total need of opioids in milligrams | Participants will be followed for the duration of post-operative hospital stay, an expected average of 7 days
Length of sick leave (days) | Participants will be followed for the duration of sick leave, depending on occupation estimated 1-4 weeks
Number of participants that develop ventral hernia | 10 years
Number of patient with recurrent adhesive small bowel obstruction | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Panu Mentula, MD, PhD, Study Director — Helsinki University Central Hospital; Ari Leppäniemi, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (8):
- Finland (6):
  - Helsinki University Central Hospital, Helsinki
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Vaasa Central Hospital, Vaasa
  - Peijas Hospital, Vantaa
- Italy (2):
  - Bologna Maggiore Hospital, Bologna
  - Parma University Hospital, Parma

REFERENCES:
- [Derived] Sallinen V, Wikstrom H, Victorzon M, Salminen P, Koivukangas V, Haukijarvi E, Enholm B, Leppaniemi A, Mentula P. Laparoscopic versus open adhesiolysis for small bowel obstruction - a multicenter, prospective, randomized, controlled trial. BMC Surg. 2014 Oct 11;14:77. doi: 10.1186/1471-2482-14-77. PMID 25306234